CLINICAL TRIAL: NCT02082132
Title: A Cross-sectional Study of Young-onset Diabetes in Two UK Ethnic Groups.
Brief Title: MODY in Young-onset Diabetes in Different Ethnicities
Acronym: MYDIABETES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 13SM0659
Record Dates: First submitted 2013-10-15; First posted 2014-03-10 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Diabetes; Maturity Onset Diabetes of the Young; Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — We will be collecting blood and urine samples for routine diabetes tests as well as more specialist tests that will help define what type of diabetes is present. We'll also collect DNA to look for MODY (maturity onset diabetes of the young), the genetic cause of diabetes, in some people.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe and compare the different types of diabetes that exist in people from white European and south Asian origin in the UK (United Kingdom) who are diagnosed with diabetes before they turn 30 years old. By doing this we hope to identify cases of MODY (maturity onset diabetes of the young), which is a rare genetic cause of diabetes that is frequently misdiagnosed. Identifying MODY cases is important, as the treatment may differ to conventional treatment for type 1 or type 2 diabetes.

DETAILED DESCRIPTION:
People who meet the recruitment criteria, will be invited to attend for a single fasted 2 hour visit at our research facility. During the visit we will record details of their diabetes history as well as their general health and undertake blood and urine tests. At the end of the visit their participation will be complete. We will contact them later to discuss results of specialist blood tests and whether or not they have MODY, if they have had genetic testing performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetes on the basis of fasting glucose and/or oral glucose tolerance test and/or HbA1c as per WHO criteria.
* Diagnosed with diabetes between 6 months and 30 years of age.
* South Asian ancestry- defined as self-reported ancestry and at least 2 grandparents from the Indian Subcontinent (India, Pakistan, Bangladesh or Sri Lanka).
* European ancestry - defined as self-reported ancestry and at least 2 grandparents from within Europe.

Exclusion Criteria:

* An established secondary cause of diabetes exists (for example recurrent pancreatitis, pancreatectomy, new onset diabetes after transplantation, Cushing's syndrome, acromegaly, steroid induced).
* Enrolled in another study.
* Have active malignancy or under investigation for malignancy.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People in the UK diagnosed with any type of diabetes before the age of 30 years from either white European or South Asian origin.
Sampling Method: Probability Sample
Enrollment: 916 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of MODY | 5 years
  Comparison of frequency of MODY mutations between two ethnic groups

SECONDARY OUTCOMES:
Comparison of biochemical and clinical characteristics in people with MODY between each ethnic group. | 5 years
  * Difference in fasting C-peptide levels between UK South Asian and white European people
  * Difference in BMI, waist and hip circumference between UK South Asian and white European people
  * Differences in affected gene between UK South Asian and white European people
Comparison of clinical and biochemical characteristics of other subtypes of diabetes | 5 years
  In people phenotyped as type 1 or type 2 diabetes:
  * Difference in fasting C-peptide levels between UK South Asian and white European people
  * Difference in BMI, waist and hip circumference between UK South Asian and white European people
  * Differences in diabetes antibody positivity between UK South Asian and white European people

CONTACTS AND LOCATIONS:
Overall Officials: Nick S Oliver, MBBS, MRCP, Study Director — Imperial College London; Shivani Misra, MBBS, MRCP, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shields BM, Hicks S, Shepherd MH, Colclough K, Hattersley AT, Ellard S. Maturity-onset diabetes of the young (MODY): how many cases are we missing? Diabetologia. 2010 Dec;53(12):2504-8. doi: 10.1007/s00125-010-1799-4. Epub 2010 May 25. PMID 20499044
- [Background] Murphy R, Ellard S, Hattersley AT. Clinical implications of a molecular genetic classification of monogenic beta-cell diabetes. Nat Clin Pract Endocrinol Metab. 2008 Apr;4(4):200-13. doi: 10.1038/ncpendmet0778. Epub 2008 Feb 26. PMID 18301398
- [Background] Porter JR, Rangasami JJ, Ellard S, Gloyn AL, Shields BM, Edwards J, Anderson JM, Shaw NJ, Hattersley AT, Frayling TM, Plunkett M, Barrett TG. Asian MODY: are we missing an important diagnosis? Diabet Med. 2006 Nov;23(11):1257-60. doi: 10.1111/j.1464-5491.2006.01958.x. PMID 17054605
- [Background] Shields BM, McDonald TJ, Ellard S, Campbell MJ, Hyde C, Hattersley AT. The development and validation of a clinical prediction model to determine the probability of MODY in patients with young-onset diabetes. Diabetologia. 2012 May;55(5):1265-72. doi: 10.1007/s00125-011-2418-8. Epub 2012 Jan 5. PMID 22218698